CLINICAL TRIAL: NCT02964923
Title: Genes Polymorphisms and Metabolic Effects of the Second Generation Antipsychotic Drugs in Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC-81571309
Record Dates: First submitted 2016-11-01; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Genetic polymorphism; Metabolic side effects of drugs; schizophrenia; Second-Generation Antipsychotic; Cannabinoid Receptor Type 1
MeSH Terms: conditions — Schizophrenia; Metabolic Side Effects of Drugs and Substances

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Olanzapine group: Following the baseline assessment, subjects will enter an open treatment group with Olanzapine(Zyprexa) lasting 6 weeks. The subjects will start with a dose of 5-10mg/d , which would be adjusted to as low as 10 mg/d or as high as 20 mg/d, based on clinical response.And drug dose adjustments must be completed within 1 week.
- Risperidone group: Following the baseline assessment, subjects will enter an open treatment group with Risperidone oral solution(Risperdal) lasting 6 weeks. The subjects will start with a dose of 1ml/d , which would be adjusted to as low as 4 ml/d or as high as 6 ml/d, based on clinical response.Drug dose adjustments interval is generally not less than 2 days, and should reach a effective dose of 4~6ml/d within 1 week.
- Ziprasidone group: Following the baseline assessment, subjects will enter an open treatment group with Ziprasidone Hydrochloride Capsules(Zeldox) lasting 6 weeks. They started with a dose of 40mg/d , which would be adjusted to as low as 80mg/d or as high as 160/d, based on clinical response.Drug dose adjustments interval is generally not less than 2 days, and should reach a effective dose of 80~160mg/d within 10 days.

SUMMARY:
The purpose of the study is to investigate these effects of Second-Generation Antipsychotic (SGAs) on glucose and lipid metabolic parameters in patients with schizophrenia, and explore the relationship between genes polymorphisms (such as drug metabolic enzyme, Endogenous Cannabinoid Receptor Type 1(CB1) and so on) and the SGAs-induced glucose and lipid metabolic disorder in Chinese Han persons with schizophrenia who are taking one of the SGAs(olanzapine, risperidone or ziprasidone).

DETAILED DESCRIPTION:
SGAs now is used as the main tool to treat schizophrenia, however，the mechanism of glucose and lipid metabolism disorder it brings is still unclear. Based on the previous studies, the investigators found that the CB1 gene has a close connection with the metabolism disorder.The investigators suppose that the CB1 also has a significant role in regulation of energy and metabolism in hypothalamus. In this study ,the investigators will recruit 300 Patients with schizophrenia who defined by Diagnostic and Statistical Manual-5 (DSM-5), aged 18 to 60,and all the participants will receive a 6-week systematic treatment by one of the SGAs(including olanzapine, risperidone oral solution, ziprasidone capsules), and a battery of assessments of treatment effect and safety. Plasma concentration will be tested regularly, and these genes polymorphisms of CB1 and other associated with energy metabolism will be conducted by the second generation of gene detection techniques.This study could provide evidence and data to achieve the aim of individualized medication, reduce the drugs' side effect, also throw light on the production of medication for correct the metabolism disorder.

ELIGIBILITY:
Inclusion Criteria:

* All cases must be in accordance with the DSM-5 schizophrenia or schizophreniform disorder diagnosis standards
* Negative and positive symptom scale(PANSS)score ≥ 60 points;Aged 18 to 60
* Did not participate diet or other body mass reduction projects
* Did not have physical illness which affects diet or activities
* Did not use any antipsychotic drug within 2 weeks
* Subject to consent by the Ethics Committee on clinical trials of drugs,Xijing hospital of The Fourth Military Medical University , all the participants signed a written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients with serious body disease, such as epilepsy, liver and kidney impairment, digestive system diseases, etc
* Obvious abnormalities on physical and laboratory examination
* Body mass index(BMI)≥25.0;Fasting plasma glucose(FPG)≥6.1mmol/L or/and 2-hour postprandial blood glucose(2hPG)≥7.8mmol/L or/and somebody has been diagnosed with diabetes and treatment;Fasting triglycerides≥2.2mmol/L
* Suffering from other mental disorders in line with DSM-5 diagnostic criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Chinese han patients with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
identification of the effect of some genes polymorphism on the development of glucose and lipid metabolism disorder in patients with schizophrenia who are treated with the SGAs | measured at week 2

SECONDARY OUTCOMES:
identification of the change of the body mass index in patients with schizophrenia who are treated with the SGAs | measured at baseline、week 2 and 6
  the ration of participants who are total remission after treatment
identification of the change of the level of Fasting Blood Sugar (FBS), 2 hours post prandial (2HPP) in patients with schizophrenia who are treated with the SGAs | measured at baseline、week 2 and 6
identification of the change of the level of lipid profile in patients with schizophrenia who are treated with the SGAs | measured at baseline、week 2 and 6
identification of the change of the level of fasting insulin in patients with schizophrenia who are treated with the SGAs | measured at baseline、week 2 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Huaning Wang, Ph.D, Study Chair — Department of Psychiatry,Xijing hospital,Xi'an,China; Zhifu Yang, Ph.D, Study Chair — Department of Pharmacy,Xijing hospital,Xi'an,China
Locations (1):
- Department of psychiatry，Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes